CLINICAL TRIAL: NCT02439840
Title: Use of Bispectral Index Monitoring to Detect Deep Sedation in Mechanically Ventilated Patients: Validity Study
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: MCS-2015-001
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Disorder; Mental, Sedative; Depressed Level of Consciousness; Mechanical Ventilation Complication; Psychosis Associated With Intensive Care
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Light sedation: Light sedation is defined as RASS of +1 to -2.
- Deep sedation: Deep sedation is defined as RASS of -3 to -5

SUMMARY:
In the previous study, the investigators obtained the cutoff value of Bispectral Index to detect early deep sedation in patients with mechanical ventilation. Bispectral Index monitoring can be used as an adjunct tool in screening and confirming deep sedation during the early period of mechanical ventilation. In present study, validation test will be carried out to clarify the sensitivity and specificity of obtained cutoff value in screening deep sedation in patients with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients are intubated and ventilated within the previous 24 hours, are administered with continuous or intermittent intravenous sedatives and/or analgesics, and are expected to receive mechanical ventilation and sedation for longer than 24 hours

Exclusion Criteria:

* Age under 18 or over 65 years;
* Continuously infusion of muscle relaxants;
* Diagnosed or suspected brain diseases, which including brain trauma, intracranial hemorrhage, stroke, brain tumors, hypoxic-ischemic encephalopathy, epilepsy and meningitis;
* Diagnosed conditions that resulted in a decrease level of consciousness, which including hypoxemia with partial pressure of oxygen in arterial blood less than 60 mmHg, hypotension with systolic blood pressure less than 90 mmHg, hypoglycemia with blood glucose concentration less than 4.1 mmol/L, anemia with hemoglobin concentration less than 70 g/L, and body temperature below 36 °C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to 3 ICUs in University Affiliated Hospital will be screened daily and enrolled consecutively.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To determine the diagnostic accuracy of BIS monitoring for detecting deep sedation against the reference standard of RASS. | 15 minutes before and after RASS evaluation
  According to RASS evaluation, observations in each time point will be stratified into 2 situations: light sedation (RASS= 0 to -2) and deep sedation (RASS= -3 to -5). Diagnostic test analysis will be applied to determine the accuracy of BIS values in predicting deep sedation.

SECONDARY OUTCOMES:
Incidence of deep sedation | 24 hours after establishing of BIS monitoring
  Number of participants with deep sedation according to RASS evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Capital Medical University
Locations (1):
- Department of Critical Care Medicine, Daxing Teaching Hospital, Capital Medical University, Beijing, Beijing Municipality, China